CLINICAL TRIAL: NCT00794235
Title: Monocentric Pilot Study Investigating the Metabolic Activity of Melanoma in Vivo During Sorafenib and Dacarbazine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Reinhard Dummer/Prof. Dr. med., Department of Dermatology, University Hospital Zurich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sorafenib and Dacarbazine
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Melanoma Stage III or IV; No Prior Chemotherapy
MeSH Terms: conditions — Melanoma | interventions — Sorafenib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib and Dacarbacine (Other)
  Interventions: Drug: Sorafenib (Nexavar), Dacarbazine (DTIC)

INTERVENTIONS:
Drug: Sorafenib (Nexavar), Dacarbazine (DTIC) — Sorafenib: 2x400 mg daily PO (2 tablets (200 mg each) each AM and PM). DAY 1-56.
  DTIC: 1-hour IV infusion 1000mg/m2 DAY 14 and 42.
  Other Names: Nexavar (Sorafenib).ATC-Code: L01XE05; Dacin (Dacarbazin).ATC-Code: L01AX04

SUMMARY:
Investigation of the metabolic activity of sorafenib and sorafenib plus dacarbazine on melanoma metastasis in patients with melanoma stage III or IV on the basis of PET/CT, LDH and S-100 evaluation. As we hypothezise a direct influence on the transcriptome by these drugs via antiproliferative or apoptotic signals, biopsies of melanoma skin metastases will be assessed with microarrays and direct changes will be revealed. If positive effects on the transcriptional profiles of metastases are revealed, patients with metastatic melanomas would benefit from these drugs resulting in tumor regressions.

Therefore, a total of 12 patients with skin- or superficial lymph node metastases with a diameter of at least 1 cm will be chosen for sorafenib therapy over 56 days per os twice daily with each 400 mg and, additionally, on day 14 and 42, intravenous dacarbazine infusion (volume depending on the body surface area (1000 mg/m2)). Before treatment with sorafenib, before treatment with dacarbazine, and after treatment, S100 and LDH will be measured in serum, PET/CT will be conducted and biopsy will be taken out of one skin metastasis on the same day.

DETAILED DESCRIPTION:
A total of 12 patients with skin- or superficial lymph node metastases with a diameter of at least 1 cm will be chosen for sorafenib therapy over 56 days per os twice daily with each 400 mg and, additionally, on day 14 and 42, intravenous dacarbazine infusion (volume depending on the body surface area (1000 mg/m2)).

On screening day, the medical history as well as the physical examination with determining the vital signs and the analyzing the coagulation status in the venous blood are conducted. In women, a pregnancy test will be conducted. On screening day, as well as on day 10, 16, 35 and 60, venous blood is taken for examination of hematology (hemoglobin, hematocrit, red blood cell (RBC) count, platelets, white blood cell (WBC) count with differential (total neutrophils, lymphocytes, monocytes, eosinophils and basophils), biochemistry (sodium, potassium, urea, creatinine, phosphate, glucose, alanine aminotransferase (ALT), gGT, alkaline phosphatase, total bilirubin, albumin, total lipid status with LDL-cholesterol, HDL-cholesterol, triglyceride), S-100, LDH, and for asservation of 40 ml EDTA and 10 ml Serum. At every consultation (screening day, day 1, 10, 14, 16, 35, 42, 60), concomitant medication will be recorded, and vital signs will be determined. At every consultation except of screening day and day 1, adverse events will be reported. FDG-PET/CT is conducted on screening day, day 10, 16 and 60; afterward, one cutaneous metastasis which was included in previous PET/CT scan, is biopsied for investigating its gene processing profile (day 60 is optional).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age > 18 years.
2. Histologically or cytologically confirmed unresectable (stage III) or metastatic (stage IV) melanoma for whom treatment with dacarbazine is considered medically acceptable.
3. No prior chemotherapy.
4. ECOG Performance Status of 0 or 1.
5. Life expectancy of at least 12 weeks.
6. Subjects with at least one uni-dimensional (for RECIST) or bi-dimensional (for WHO) measurable lesion. Lesions must be measured by CT-scan or MRI.
7. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening: Hemoglobin >= 9.0 g/dl. Absolute neutrophil count (ANC) >=1,500/mm3. Platelet count >=100,000/ìl. Total bilirubin <= 1.5 times the upper limit of normal. ALT and AST <= 2.5 x upper limit of normal (< 5 x upper limit of normal for patients with liver involvement of their cancer). Alkaline phosphatase < 4 x ULN. PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists]. Serum creatinine <= 1.5 x upper limit of normal.
8. Signed and dated informed consent before the start of specific protocol procedures.
9. Baseline serum LDH level > 1.1 ULN.
10. Assessable metastases (Skin or superficial lymph nodes, minimal diameter 1 cm)

EXCLUSION CRITERIA:

1. History of cardiac disease: congestive heart failure > NYHA class
2. active CAD (MI more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
3. History of HIV infection or chronic hepatitis B or C.
4. Active clinically serious infections (> grade 2 NCI-CTC version 3.0).
5. Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry).
6. Patients with seizure disorder requiring medication (such as steroids or anti-epileptics).
7. History of organ allograft.
8. Patients with evidence or history of bleeding diathesis.
9. Patients undergoing renal dialysis.
10. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
11. Primary ocular melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
1) Metabolic activity (glucose-uptake) in vivo, standardised uptake value (SUV) in FDG-PET/CT. 2) Quantification of soluble S100 serum and LDH. 3) Gene expression profile of cutaneous melanoma metastasis | SCREEN: S100, LDH, FDG-PET/CT, biopsy. DAY10: S100, LDH, FDG-PET/CT, biopsy. DAY16: S100, LDH, FDG-PET/CT, biopsy. DAY35: S100, LDH. DAY60: S100, LDH, FDG-PET/CT, biopsy (biopsy is optional). Sorafenib: DAY1-56. DTIC: DAY 14 and 42.

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Dummer, MD, Principal Investigator — Department of Dermatology, University Hospital Zurich, Switzerland
Locations (1):
- Department of Dermatology, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland